CLINICAL TRIAL: NCT06855056
Title: Validation of New Prognostic biomarkerRs in Patients With cirrhOsis diScharged After a hosPitalization Due to acutE deCompensation or acuTe-on-chronic Liver Failure
Brief Title: Validation of New Prognostic Biomarkers in Patients With Decompensated Cirrhosis
Acronym: PROSPECT
Status: Recruiting | Type: Observational
Sponsor: European Foundation for Study of Chronic Liver Failure (Other)
Collaborators: Universität Münster (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Hospital Universitari Vall d'Hebron Research Institute (Other); Hospital Clinic de Barcelona, Barcelona, Spain (Unknown); Hospital Universitario Ramon y Cajal (Other); Beaujon Hospital (Other); University Hospital, Aachen (Other); A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Other Study IDs: PROSPECT; 847949 (Other Grant/Funding Number: European Health and Digital Executive Agency)
Record Dates: First submitted 2025-02-10; First posted 2025-03-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Liver Cirrhosis; Decompensated Cirrhosis of Liver
Keywords: Decompensated Liver Cirrhosis; Acute on Chronic Liver Failure (ACLF); Liver Diseases; Liver Cirrhosis; Biomarkers
MeSH Terms: conditions — Liver Cirrhosis; Acute-On-Chronic Liver Failure; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Decompensated Liver Cirrhosis: Patients eligible for this study will be patients with decompensated cirrhosis expected to be discharged from the hospital within 48 hours after an index admission for AD according to the EASL-CLIF criteria

SUMMARY:
The study aims to test the effectiveness of new biomarkers (measurable molecules in our body) in predicting the health outcome of patients with liver cirrhosis discharged from the hospital after a serious complication of the disease

DETAILED DESCRIPTION:
The PROSPECT study is part of the larger EU H2020 DECISION project, which aims to analyze and clarify the pathophysiological mechanisms of decompensated cirrhosis at the systemic level and its transition to ACLF, with the goal of significantly reducing mortality through therapies tailored to the specific needs of individual patients or patient groups.

As planned in the DECISION project, the biological samples of three large cohorts of patients with cirrhosis admitted to hospital for acute decompensation (AD) without ACLF, deriving from the EF-CLIF-promoted observational studies CANONIC and PREDICT (Europe) and ACLARA (South America) were analyzed to measure lipidomics, epigenomics, whole-blood transcriptomics, micro-RNA, serum metabolomics, plasma cytokines, and plasma extracellular vesicles.

Both system medicine approaches and more traditional methods of analysis have been applied to analyze and interpret the results. The analyses are still ongoing due to the very high number of variables and the complexity of associating -omics to clinical data, yet, some of these analyses have already generated solid data allowing the identification of novel biomarkers which can be further tested.

In the PROSPECT study, patients hospitalized for acute decompensation of liver cirrhosis, who meet the inclusion and exclusion criteria, will be enrolled after providing signed informed consent. Participants will be screened and included in the study within 48 hours prior to the expected discharge from the hospital. The study will last 180 days and will include an initial visit during which clinical parameters and additional blood samples will be collected, followed by two follow-up visits - which can also be conducted by phone - during which only clinical information will be gathered. Samples will be analyzed to determine the biomarkers selected within the DECISION project and parameters related to the following pathophysiological mechanisms:

* systemic inflammation
* blood and microRNA transcriptome
* the metabolomic landscape
* albumin structure and function
* coagulation assays
* extracellular vesicles
* endothelial function

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Patients with decompensated cirrhosis admitted to hospital due to AD according to the EASL-CLIF criteria (rapid onset of ascites, hepatic encephalopathy, portal hypertensive- related gastrointestinal bleeding, bacterial infection, or any combination of these), including those who presented ACLF during hospitalization.
3. Recovery from AD and expected to be discharged within the next 48 hours.

Exclusion Criteria:

1. Admission for planned diagnostic or therapeutic procedures
2. Active malignancy (except for hepatocellular carcinoma within the Milan criteria or nonmelanocytic skin cancer)
3. Antiviral treatment for hepatitis C, B and delta initiated in the last 6 months or planned to be initiated in the following 6 months.
4. HIV positive (except undergoing treatment and who do not exhibit clinical manifestations of AIDS).
5. Ongoing alcohol use disorder with an expected low adherence to prescriptions as judged by physician
6. Previous liver or other organ transplantation
7. Patients with TIPS or other surgical porto-caval shunts
8. Chronic organic renal failure stage IV and V or estimated Glomerular Filtration Rate <20 ml/min according to the MDRD equations
9. Chronic heart failure NYHA class III or IV
10. Pulmonary disease GOLD III or IV
11. Patients with a history of significant extrahepatic disease with life expectancy <6 months
12. Severe psychiatric disorders
13. Pregnancy and breast-feeding
14. Expected low adherence to study protocol as judged by physician
15. Patients who cannot provide written informed consent or refuse to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for this study will be patients with decompensated cirrhosis expected to be discharged from the hospital within 48 hours after an index admission for AD according to the EASL-CLIF criteria.
Sampling Method: Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To test the prognostic accuracy of novel biomarkers identified within the DECISION project. | Until September 30th 2025
  The primary objective will be evaluated assessing the following end-point:
  ● Survival at 3 months

SECONDARY OUTCOMES:
To characterize the clinical and biological features at the time of discharge predicting the 6-month outcome and the different trajectories of patients surviving a hospitalization for AD complicated or not by ACLF. | Until September 30th 2025
  Secondary objectives will be evaluated assessing the following end-points:
  * Survival at 6 months
  * Incidence of emergent re-admissions to hospital at 3 months due to liver related causes
  * Incidence of emergent re-admissions to hospital at 6 months due to liver related causes
  * Incidence of emergent re-admissions to hospital at 3 months due to non liver related causes
  * Incidence of emergent re-admissions to hospital at 6 months due to non liver related causes
  * Incidence of ACLF at 3 months
  * Incidence of ACLF at 6 months
  * Incidence of TIPS insertion at 3 months
  * Incidence of TIPS insertion at 6 months

CONTACTS AND LOCATIONS:
Locations (9):
- Hospital Beaujon, Clichy, France, France
- Germany (2):
  - University Hospital, Aachen, Aachen, Germany
  - Universitätsklinikum Münster, Münster, Germany
- Italy (2):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico di S.Orsola, Bologna, Italia
  - A.O.U. Città della Salute e della Scienza di Torino, Torino, Italy
- Spain (3):
  - Hospital Universitari Vall d'Hebron Research Institute, Barcelona, Spain
  - Hospital Clinic de Barcelona, Barcelona, Spain
  - Hospital Universitario Ramon y Cajal, Madrid, Spain
- Royal Free Hospital, London, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: No